CLINICAL TRIAL: NCT02180165
Title: A Randomized, Comparative, Open-label Study to Assess the Safety and Efficacy of MK-5592 Compared With Voriconazole in Japanese Subjects With Deep-seated Fungal Infection
Brief Title: Assessing the Safety and Efficacy of MK-5592 (Posaconazole) in Japanese Participants With Fungal Infection (MK-5592-101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5592-101; 142639 (Registry Identifier: JAPIC-CTI); MK-5592-101 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — posaconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: Posaconazole (Experimental): 300 mg posaconazole oral tablet (or 300 mg intravenous (IV) solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
  Interventions: Drug: Posaconazole
- Cohort 1: Voriconazole (Active Comparator): 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
  Interventions: Drug: Voriconazole
- Cohort 2: Posaconazole (Experimental): 300 mg posaconazole oral tablet (or 300 mg intravenous (IV) solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
  Interventions: Drug: Posaconazole
- Cohort 2: Voriconazole (Active Comparator): 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Posaconazole — 300 mg posaconazole twice on Day 1, either by oral tablet or IV solution; followed by 300 mg once daily for up to 84 days
  Arms: Cohort 1: Posaconazole; Cohort 2: Posaconazole
Drug: Voriconazole — 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
  Arms: Cohort 1: Voriconazole; Cohort 2: Voriconazole

SUMMARY:
The primary objective of this study is to assess and compare the safety of posaconazole with voriconazole in Japanese participants with aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=45 kg
* Can be treated by taking tablet orally or intravenous (IV) formulation via central vein
* Female has a negative pregnancy test
* Female of non-childbearing potential; or if of childbearing potential, agrees to use proper combination of barrier method of birth control
* Met screening criteria for either Invasive aspergillosis, chronic pulmonary aspergillosis, zygomycosis or fusariosis.

Exclusion Criteria:

* Has a fungal infection other than Aspergillus any species (spp.) Zygomycetes (including Mucor spp.) and Fusarium spp. infection
* Has allergic bronchopulmonary aspergillosis, allergic sinusitis of aspergillosis, or aspergillosis of the eye
* Has long-term inactive aspergilloma not expected to respond to investigational product
* Is not expected to survive study duration
* Has an underlying disease, complication and systemic condition which makes it difficult to evaluate effect of study drug
* Has received, or continues to receive any systemic antifungal therapy, and cannot discontinue this treatment; but if fungal infection does not improve, can switch to study drug
* Is expected to need prohibited medications
* Has received posaconazole, has received voriconazole for this infection in the past and has deep-seated fungal infection that has not responded to this treatment, has intolerance for azole antifungal treatments, or is receiving antifungal combination therapy for chronic pulmonary aspergillosis
* Has known hypersensitivity to any medication
* Has history of either Torsade de Pointes, myocardial infarction within previous 90 days, has congenital or acquired long QT interval syndrome, or unstable cardiac arrhythmia
* Has significant liver dysfunction
* Has liver cirrhosis or cholestasis
* Has renal insufficiency
* Has a known hereditary problem of either galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Has acute symptomatic pancreatitis within 6 months of study entry or chronic pancreatitis
* Has an active skin lesion consistent with squamous cell carcinoma or melanoma, or within prior 5 years a history of malignant melanoma
* Has known or suspected Gilbert's disease
* Female is pregnant, or nursing, or intends to become pregnant within 14 days after end of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] "Kohno S, Izumikawa K, Yoshida M, Okada F, Mori T, Najima Y, Waskin H, Shizuya T, Fukuhara T, Adachi N, Niki Y. A Randomized, Active-controlled, Open-label, Comparative Study to Assess the Safety and Efficacy of Posaconazole in Japanese Subjects with Deep-seated Fungal Infection. Nihon Ishinkin Gakkai Zasshi. 2020; 61(1):1-11. PDF file: https://www.jstage.jst.go.jp/article/ishinkin/61/1/61_19-00015/_pdf/-char/ja Web page: https://www.jstage.jst.go.jp/article/ishinkin/61/1/61_19-00015/_article/-char/ja"

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in male and female Japanese participants with deep-seated fungal infection.
Groups:
- Cohort 1: Posaconazole: Participants with chronic pulmonary aspergillosis or with fusariosis or zygomycosis, received 300 mg posaconazole oral tablet (or 300 mg intravenous [IV] solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 1: Voriconazole: Participants with chronic pulmonary aspergillosis received 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
- Cohort 2: Posaconazole: Participants with aspergillosis or with fusariosis or zygomycosis received 300 mg posaconazole oral tablet (or 300 mg IV solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Voriconazole: Participants with aspergillosis received 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
Period: Overall Study
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Started (Randomized participants) | 15 | 7 | 63 | 31
Treated Participants | 15 | 7 | 62 | 31
Type of Aspergillosis | 15 (Chronic Pulmonary Aspergillosis) | 7 (Chronic Pulmonary Aspergillosis) | 57 (Invasive Aspergillosis and Chronic Pulmonary Aspergillosis) | 27 (Invasive Aspergillosis and Chronic Pulmonary Aspergillosis)
Completed (Completed Through Day 84) | 4 | 6 | 34 | 25
Not Completed | 11 | 1 | 29 | 6
Not completed — Not Treated | 0 | 0 | 1 | 0
Not completed — Adverse Event | 7 | 0 | 18 | 3
Not completed — Lack of Efficacy | 0 | 1 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Cohort 1: All randomized and treated participants with chronic pulmonary aspergillosis; Cohort 2: All randomized and treated participants with invasive aspergillosis and chronic pulmonary aspergillosis
Groups:
- Cohort 1: Posaconazole: Participants with chronic pulmonary aspergillosis received 300 mg posaconazole oral tablet (or 300 mg intravenous (IV) solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Posaconazole: Participants from cohort 2 with invasive aspergillosis and chronic pulmonary aspergillosis received 300 mg posaconazole oral tablet (or 300 mg IV solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Voriconazole: Participants from cohort 2 with invasive aspergillosis and chronic pulmonary aspergillosis received 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole | Total
Number analyzed (Participants) | 15 | 7 | 57 | 27 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.5) | 69.9 (4.5) | 65.6 (12.3) | 58.2 (13.9) | 63.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 12 | 4 | 54 | 25 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 7 | 57 | 27 | 106
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: Up to approximately Day 98
Population: Cohort 1: All randomized participants with chronic pulmonary aspergillosis who received at least one dose of study treatment. Cohort 2: All randomized participants with invasive aspergillosis and chronic pulmonary aspergillosis who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Posaconazole: Participants with chronic pulmonary aspergillosis received 300 mg posaconazole oral tablet (or 300 mg IV solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Posaconazole: Participants from cohort 2 with invasive and chronic pulmonary aspergillosis received 300 mg posaconazole oral tablet (or 300 mg IV solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Voriconazole: Participants from cohort 2 with invasive and chronic pulmonary aspergillosis received 300 mg voriconazole oral tablet (or 6 mg/kg IV solution) twice on Day 1, followed by 200 mg oral tablet (or 4 mg/kg IV solution) twice daily for up to 84 days
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 15 | 7 | 57 | 27
Participants | 15 | 6 | 57 | 27

2. Secondary Outcome: Percentage of Participants With Successful Overall Response for Invasive Aspergillosis in Cohort 2 at Day 42
Description: Successful treatment (or successful overall response) is defined as complete response and partial response to treatment assessed by the clinical adjudication committee (CAC). The 95% confidence interval (CI) is based on the Clopper-Pearson exact method.
Time Frame: Day 42
Population: Participants in cohort 2 diagnosed by CAC with proven or probable invasive aspergillosis; who received at least one dose of study treatment; and had a baseline observation for the analysis endpoint. Participants in cohort 1 were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants |  |  | 40.0 [5.3 to 85.3] | 100 [29.2 to 100]

3. Secondary Outcome: Percentage of Participants With Successful Overall Response for Invasive Aspergillosis in Cohort 2 at Day 84
Description: Successful treatment (or successful overall response) is defined as complete response and partial response to treatment assessed by CAC. The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 84
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants |  |  | 60.0 [14.7 to 94.7] | 100 [29.2 to 100]

4. Secondary Outcome: Percentage of Participants With Successful Overall Response for Chronic Pulmonary Aspergillosis in Cohort 2 at Day 42
Description: Successful treatment (or successful overall response) is defined as favorable response to treatment assessed by CAC. The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 42
Population: Participants in cohort 2 diagnosed by CAC with proven or probable chronic pulmonary aspergillosis; who received at least one dose of study treatment; and had a baseline observation for the analysis endpoint. Participants in cohort 1 were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 56.3 [41.2 to 70.5] | 87.0 [66.4 to 97.2]

5. Secondary Outcome: Percentage of Participants With Successful Overall Response for Chronic Pulmonary Aspergillosis in Cohort 2 at Day 84
Description: as for outcome 4
Time Frame: Day 84
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 58.3 [43.2 to 72.4] | 87.0 [66.4 to 97.2]

6. Secondary Outcome: Percentage of Participants With Successful Overall Response for Invasive Aspergillosis and Chronic Pulmonary Aspergillosis in Cohort 2 at End of Trial (Day 84)
Description: Successful treatment (or successful overall response) for invasive aspergillosis is defined as complete response and partial response to treatment assessed by CAC. Successful treatment (or successful overall response) for chronic pulmonary aspergillosis is defined as favorable response to treatment.The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 84
Population: Participants in cohort 2 diagnosed by CAC with proven or probable invasive aspergillosis or chronic pulmonary aspergillosis; who received at least one dose of study treatment; and had a baseline observation for the analysis endpoint. Participants in cohort 1 were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 53 | 26
Percentage of participants |  |  | 58.5 [44.1 to 71.9] | 88.5 [69.8 to 97.6]

7. Secondary Outcome: Percentage of Participants With Successful Overall Response for Zygomycosis in Cohort 2 at Day 42
Description: Zygomycosis is an infection caused by zygomycete fungi. Successful treatment (or successful overall response) is defined as complete response and partial response to treatment assessed by CAC. The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 42
Population: Participants in cohort 2, posaconazole treatment only, diagnosed by CAC with proven or probable zygomycosis; who received at least one dose of study treatment; and had a baseline observation for the analysis endpoint. Participants in cohort 1, and cohort 2 voriconazole treatment were not analyzed for this outcome measure.
Measure: Number; unit: Percentage of participants
Groups:
- Cohort 2: Posaconazole: Participants from cohort 2 with zygomycosis received 300 mg posaconazole oral tablet (or 300 mg IV solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 3 | 0
Percentage of participants |  |  | 66.7 |

8. Secondary Outcome: Percentage of Participants With Successful Overall Response for Zygomycosis in Cohort 2 at Day 84
Description: as for outcome 7
Time Frame: Day 84
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 3 | 0
Percentage of participants |  |  | 100 |

9. Secondary Outcome: Percentage of Participants With Successful Overall Response for Invasive Aspergillosis in Cohort 2 at Day 42 as Assessed by the Clinical Investigator
Description: Successful treatment (or successful overall response) for invasive aspergillosis is defined as complete response and partial response to treatment assessed by the clinical investigator.The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants |  |  | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2]

10. Secondary Outcome: Percentage of Participants With Successful Overall Response for Chronic Pulmonary Aspergillosis in Cohort 2 at Day 84 as Assessed by the Clinical Investigator
Description: Successful treatment (or successful overall response) for chronic pulmonary aspergillosis is defined as favorable response to treatment assessed by the clinical investigator.The 95% CI is based on the Clopper-Pearson exact method.
Time Frame: Day 84
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 60.4 [45.3 to 74.2] | 78.3 [56.3 to 92.5]

11. Secondary Outcome: Percentage of Participants With Invasive Aspergillosis With Clinical Response of Resolution or Improvement in Cohort 2 at Day 42
Description: A clinical response of resolution is defined as resolution of attributable signs and symptoms of disease, and a clinical response of improvement is defined as improvement of attributable signs and symptoms of disease as assessed by the CAC.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants
  Resolution |  |  | 60.0 | 0
  Improvement |  |  | 20.0 | 66.7

12. Secondary Outcome: Percentage of Participants With Invasive Aspergillosis With Clinical Response of Resolution or Improvement in Cohort 2 at Day 84
Description: as for outcome 11
Time Frame: Day 84
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants
  Resolution |  |  | 60.0 | 33.3
  Improvement |  |  | 20.0 | 33.3

13. Secondary Outcome: Percentage of Participants With Invasive Aspergillosis With Radiological Response of Resolution or Improvement in Cohort 2 at Day 42
Description: A radiological response of resolution is defined as resolution of radiological lesions, and a radiological response of improvement is defined as major reduction in size of radiological lesions as assessed by the CAC.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants
  Resolution |  |  | 0 | 0
  Improvement |  |  | 40.0 | 100

14. Secondary Outcome: Percentage of Participants With Invasive Aspergillosis With Radiological Response of Resolution or Improvement in Cohort 2 at Day 84
Description: as for outcome 13
Time Frame: Day 84
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants
  Resolution |  |  | 0 | 0
  Improvement |  |  | 60.0 | 100

15. Secondary Outcome: Percentage of Participants With Invasive Aspergillosis With Mycological Response of Eradication in Cohort 2 at Day 42
Description: A mycological response of eradication is defined as fungus detected from culture or microscopy at the screening is eradicated at the time of evaluation (including presumed eradication), as assessed by the CAC.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 5 | 3
Percentage of participants |  |  | 20.0 | 0

16. Secondary Outcome: Percentage of Participants With Chronic Pulmonary Aspergillosis With Clinical Response of Resolution in Cohort 2 at Day 42
Description: A clinical response of resolution is defined as resolution of attributable signs and symptoms of disease, as assessed by the CAC.
Time Frame: Day 42
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 43.8 | 73.9

17. Secondary Outcome: Percentage of Participants With Chronic Pulmonary Aspergillosis With Clinical Response of Resolution in Cohort 2 at Day 84
Description: as for outcome 16
Time Frame: Day 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 45.8 | 82.6

18. Secondary Outcome: Percentage of Participants With Chronic Pulmonary Aspergillosis With Radiological Response of Resolution in Cohort 2 at Day 42
Description: A radiological response of resolution is defined as resolution of radiological lesions, as assessed by the CAC.
Time Frame: Day 42
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 58.3 | 87.0

19. Secondary Outcome: Percentage of Participants With Chronic Pulmonary Aspergillosis With Mycological Response of Eradication in Cohort 2 at Day 42
Description: as for outcome 15
Time Frame: Day 42
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 33.3 | 21.7

20. Secondary Outcome: Percentage of Participants With Chronic Pulmonary Aspergillosis With Mycological Response of Eradication in Cohort 2 at Day 84
Description: as for outcome 15
Time Frame: Day 84
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
Number analyzed (Participants) | 0 | 0 | 48 | 23
Percentage of participants |  |  | 35.4 | 21.7

ADVERSE EVENTS:
Time Frame: Up to approximately Day 98
Description: All randomized participants who received at least one dose of study treatment.
Groups:
- Cohort 1: Posaconazole: Participants with chronic pulmonary aspergillosis or with fusariosis or zygomycosis, received 300 mg posaconazole oral tablet (or 300 mg intravenous (IV) solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days
- Cohort 2: Posaconazole: Participants with aspergillosis or with fusariosis or zygomycosis,received 300 mg posaconazole oral tablet (or 300 mg intravenous (IV) solution) twice on Day 1, followed by 300 mg oral tablet or IV solution once daily for up to 84 days. Participants with fusariosis or zygomycosis, were also assigned to this treatment group
Arm/Group | Cohort 1: Posaconazole | Cohort 1: Voriconazole | Cohort 2: Posaconazole | Cohort 2: Voriconazole
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/7 | 6/62 | 0/31
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/7 | 28/62 | 3/31
Other Adverse Events (participants affected / at risk) | 15/15 | 6/7 | 58/62 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Posaconazole (N=15) | Cohort 1: Voriconazole (N=7) | Cohort 2: Posaconazole (N=62) | Cohort 2: Voriconazole (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blister infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 7 (7) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Posaconazole (N=15) | Cohort 1: Voriconazole (N=7) | Cohort 2: Posaconazole (N=62) | Cohort 2: Voriconazole (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colour blindness acquired (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 2 (2) | 5 (5) | 9 (9)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 11 (12) | 5 (5)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 5 (6) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 0 (0) | 18 (19) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 13 (14) | 6 (6)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (2) | 1 (2) | 4 (6)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 7 (7) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 8 (8) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 4 (4) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 3 (4) | 1 (1)
Blood potassium decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 6 (6) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 2 (3)
Renal function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 10 (11) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 13 (13) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT02180165/Prot_SAP_000.pdf